CLINICAL TRIAL: NCT05644327
Title: The Effects of Different Exercise Modalities on Sleep Quality and Architecture in People With Parkinson's Disease
Brief Title: Exercise to Improve Sleep in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Jewish Rehabilitation Hospital (Other); The Memory Lab (Unknown); The Human Brain Control of Locomotion Lab (HBCL) (Unknown); The Cummings Centre (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marc Roig, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP5020221584
Record Dates: First submitted 2022-11-18; First posted 2022-12-09 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Rehabilitation; Sleep; Exercise; Cardiovascular training; Resistance training; Multimodal training; Motor function; Cognition; Quality of life
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Assessors will be blinded to the participants' group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cardiovascular training (CT) (Experimental): Cardiovascular training (CT) will be performed on a recumbent stepper. CT will start at low intensity, and, through a linear progression, will reach vigorous intensity; then, this intensity will be maintained until the end of the training period. Each session will include five minutes of warm-up and cool-down performed at the beginning and at the end of the training, respectively. Furthermore, five minutes of stretching will be performed after the cool-down. CT's sessions will last approximately 45 minutes (30 to 50 minutes) and will be interspersed with 48 hours of recovery.
  Interventions: Behavioral: Cardiovascular training (CT)
- Resistance training (RT) (Experimental): Resistance training (RT) intensity will be estimated using the percentage of one-maximal repetition (1-RM) defined as the maximal weight liftable for ten maximal repetitions with proper form. The program will include five exercises (leg press, lat machine, leg extension, leg curl, bench press) and will start at high-volume low intensity. RT will follow a periodization to reach high-intensity low-volume at the end of the intervention (week 12). The training sessions will start and end with five-minute of warm-up and cool-down, which will include exercise on a recumbent stepper and stretching, respectively. RT's sessions will last approximately 45 minutes (40 to 50 minutes) and will be interspersed with 48 hours of recovery.
  Interventions: Behavioral: Resistance training (RT)
- Multimodal training (MT) (Experimental): Multimodal training (MT) will combine cardiovascular and resistance training interventions using the modalities described previously, but each component will be shortened to match the overall training duration (i.e., volume) among groups. The first part of each training session will always include three resistance exercises, which will be followed by 15-20 minutes of cardiovascular training performed on the total body recumbent stepper. Periodization will follow the same progression previously described for cardiovascular and resistance training, respectively, reaching vigorous intensity towards the end of the training period. Training sessions will include a five-minute warm-up and cool-down on the total body recumbent stepper. MT's sessions will approximately last 45 minutes (40 to 50 minutes) and will be interspersed with 48 hours of recovery.
  Interventions: Behavioral: Multimodal training (MT)
- Control condition (CON; waiting list) (No Intervention): The control condition (CON; waiting list) will receive no intervention (i.e., exercise) but usual care. Participants in the CON will be required to go about their normal life, maintaining their current physical activity levels until the end of the study. Then, they will be offered to join one of the training programs/condition.

INTERVENTIONS:
Behavioral: Cardiovascular training (CT) — 12 weeks of CT
  Arms: Cardiovascular training (CT)
Behavioral: Resistance training (RT) — 12 weeks of RT
  Arms: Resistance training (RT)
Behavioral: Multimodal training (MT) — 12 weeks of MT
  Arms: Multimodal training (MT)

SUMMARY:
This study will investigate the impact of three common exercise modalities, cardiovascular, resistance, and multimodal (i.e., a combination of the previous two) training, on sleep quality and architecture in persons with Parkinson's disease (PD). Furthermore, the project will investigate whether the potential positive exercise-induced changes in sleep are associated with improvements in different quality of life (QoL)-related aspects. Participants will perform either cardiovascular training (CT), resistance training (RT), multimodal training (MT), or will be allocated to a control condition (i.e., waiting list - CON) for 12 weeks. Training will be performed three times/week. The assessments will be conducted at baseline, post-intervention, and follow-up (i.e. 8 weeks after the intervention) by assessors blinded to the participants' group allocation.

DETAILED DESCRIPTION:
Background: Over 100,000 Canadians are currently living with PD. Every year, 6,600 new cases are diagnosed and this number is expected to double by 2031. Almost all (98%) of those persons experience sleep problems, which can appear even before the onset of the cardinal motor symptoms of the disease, affecting multiple aspects of their QoL. Persons with PD also show alterations in sleep architecture, which are clinically relevant as they have been associated with a faster disease progression. Since medications used to reduce sleep problems in PD have potential adverse side effects, exercise has been proposed as a potential non-pharmacological alternative to improve sleep quality and architecture in people with PD. However, the most beneficial intervention to improve sleep in this clinical population is still to be determined.

Objective: 1) To conduct a 12-week RCT comparing the effects of CT, RT, MT, and CON on both objective and subjective measures of sleep quality and architecture in patients with mild-to-moderate PD; 2) To assess whether, regardless of the exercise modality, positive changes in sleep quality and architecture mediate exercise-induced improvements in aspects directly related to QoL such as cognitive and motor function.

Design: A four-arm, parallel-group, multi-site, single-blinded RCT with assessments performed at baseline (T0) and after 12 weeks of training (T1), as well as at 8 weeks post-intervention (T2), by assessors blinded to the participants' group allocation.

Methods: After completing T0, participants will be randomly allocated into four groups using a sequence created and held by a central randomization service (https://www.randomizer.at) using a 1:1:1:1 ratio. Permuted blocks of varying sizes to ensure balance over time will be used. Adherence to the training programs and training intensity progression will be monitored by trainers who will track attendance and record responses to exercise (e.g., HR) during training sessions. Participants who will miss training sessions due to valid reasons (e.g., doctor appointments) will be offered make-up sessions to complete the full 36 training sessions. Participants who do not complete 80% of the training (>27 training sessions) over the 12-week, develop injuries that preclude safety during training, or desire to stop the program, will be excluded.

Changes in objective and subjective measures of sleep quality will be assessed with polysomnography and the PD sleep scale version 2, respectively. Sleep architecture will be measured with polysomnography. Motor and cognitive function will be assessed with the Unified PD Rating Scale part III and the Scale for Outcomes in PD-Cognition, respectively. Fatigue, psychosocial functioning and QoL will be assessed with the PD Fatigue Scale, the Scale for Outcomes in PD-Psychosocial and the PD QoL Scale, respectively. The plasma concentration of different inflammatory biomarkers will be assessed using enzyme-linked immunosorbent assays (ELISA) kits following the instructions provided by the manufacturers. Cardiorespiratory fitness will be assessed with a graded exercise test (GXT) performed on a recumbent stepper.

Expected results: 1) MT will be more effective than RT, CT, and CON at improving objective and subjective sleep quality and sleep architecture; 2) Sleep architecture improvements, regardless of the type of exercise performed, will mediate enhancements in cognition and motor function; 3) Improvements in sleep quality (i.e., sleep efficiency), regardless of the type of exercise performed, will mediate enhancements in different QoL-related aspects such as fatigue and psychological functioning.

Impact: This will be the first study comparing the effect of MT, CT and RT on sleep quality and architecture and investigating whether these changes mediate improvements in cognitive and motor function as well as QoL-related aspects (e.g., fatigue). The results of the study will provide important information to design more personalized exercise-based treatments, which are patient-oriented and aimed at optimizing the effect of sleep on cognitive and motor function as well as QoL in PD.

ELIGIBILITY:
Inclusion Criteria:

* Persons with mild-moderate idiopathic Parkinson's Disease (Modified Hoehn & Yahr Scale stages 0.5-3.5);
* On a stable dosage of medication during the previous month;
* Having poor sleep quality defined as a score > 15 in the PDSS-2;

Exclusion Criteria:

* Having atypical parkinsonism, dementia, stroke, or any other neurological condition;
* Presenting severe untreated obstructive sleep apnea (OSA);
* Having a Montreal Cognitive Assessment (MoCA) score <18
* Having a Beck Depression Inventory score >31;
* Having absolute contraindications to exercise;
* Having severe osteoporosis;
* Participating in an exercise or drug trial during the period of the study;
* Exceeding the physical activity levels recommended for the general population (≥150 minutes/week of moderate-intensity or ≥75 minutes/week of vigorous-intensity cardiovascular activity) and/or strengthening activities ≥2 days/week.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in objective sleep quality | 12 weeks (post-intervention) and 8 weeks (follow-up)
  Sleep efficiency (SE) measured with polysomnography; SE (%) = Time asleep while in bed * 100; values = 0-100%; higher values reflect better SE.
Changes in subjective sleep quality | 12 weeks (post-intervention) and 8 weeks (follow-up)
  PD Sleep Scale version 2 (PDSS-2); values = 0-60; higher values reflect worse sleep quality.
Changes in sleep architectures | 12 weeks (post-intervention) and 8 weeks (follow-up)
  Changes in slow-wave power measured with polysomnography.
Changes in sleep architectures | 12 weeks (post-intervention) and 8 weeks (follow-up)
  Changes in sleep spindles density measured with polysomnography.
Changes in sleep architectures | 12 weeks (post-intervention) and 8 weeks (follow-up)
  Changes in REM sleep duration (%) measured with polysomnography.

SECONDARY OUTCOMES:
Changes in motor function | 12 weeks (post-intervention) and 8 weeks (follow-up)
  Unified PD Rating Scale part III (UPDRS part III); values = 0-132; higher values reflect worse motor function.
Changes in cognitive function | 12 weeks (post-intervention) and 8 weeks (follow-up)
  Scale for Outcomes in PD-Cognition (SCOPA-COG); values = 0-43; higher values reflect better cognitive function.
Changes in fatigue | 12 weeks (post-intervention) and 8 weeks (follow-up)
  PD Fatigue Scale; values = 16-80; higher values reflect worse fatigue.
Changes in psychosocial functioning | 12 weeks (post-intervention) and 8 weeks (follow-up)
  Scale for Outcomes in PD-Psychosocial (SCOPA-PS); values = 0-100%; higher values (%) reflect worse psychosocial functioning.
Changes in Quality of Life Scale | 12 weeks (post-intervention) and 8 weeks (follow-up)
  PD Quality of Life Scale (PDQUALIF); values = 0-100%; higher values (%) reflect worse quality of life.

OTHER OUTCOMES:
Inflammatory biomarkers | 12 weeks (post-intervention) and 8 weeks (follow-up)
  peripheral concertation of pro-inflammatory blood biomarkers (e.g., IL-6, Il-1, TNF-α); values of pro-inflammatory blood biomarkers will be reported as pg/ml.
Cardiorespiratory fitness | 12 weeks (post-intervention) and 8 weeks (follow-up)
  VO2 peak measured during a Graded Exercise Test (GXT)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Roig, Ph.D., Principal Investigator — McGill University
Locations (3):
- Canada (3):
  - Jewish Rehabilitation Hospital, Laval, Quebec
  - Human Brain Control of Locomotion Laboratory, Montreal, Quebec
  - Cummings Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No